CLINICAL TRIAL: NCT01635894
Title: A Community Intervention Study of Female Pelvic Floor Condition and Knowledge of Pelvic Floor Exercises
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Plymouth NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1706; WellBeing of Women (Other Grant/Funding Number: PG428/02)
Record Dates: First submitted 2012-07-03; First posted 2012-07-10 (Estimated); Last update posted 2015-11-05 (Estimated); Status verified 2015-11

CONDITIONS: Behavioural
Keywords: female pelvic floor condition; pelvic floor training; supervised pelvic floor training; practice nurse; nurse specialist

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- nurse specialist (Experimental): Women were screened for a "weak pelvic floor" (modified Oxford score, MOS, ≤ 2) before being invited into the trial. The women were seen monthly after their initial assessment and training and were followed-up for their final assessment at 3 months.
  Interventions: Behavioral: Training
- practice nurse (Experimental): Women were screened for a "weak pelvic floor" (modified Oxford score, MOS, ≤ 2) before being invited into the trial. The women were seen monthly after their initial assessment and training and were followed-up for their final assessment at 3 months.
  Interventions: Behavioral: Training
- Control (No Intervention): Women were screened for a "weak pelvic floor" (modified Oxford score, MOS, ≤ 2) before being invited into the trial. The women were seen monthly after their initial assessment (but no training given) and were followed-up for their final assessment at 3 months.

INTERVENTIONS:
Behavioral: Training — Women in both the practice nurse and specialist nurse groups were given supervised pelvic floor exercise training. After the initial training they were given a daily exercise regimen and seen at monthly intervals for three months. The practice nurses had attended a study day on supervising Pelvic Floor Muscle Training(PFMT)followed by practice sessions with patients overseen by the nurse specialist.
  Other Names: Pelvic Floor Muscle Training (PFMT)
  Arms: nurse specialist; practice nurse

SUMMARY:
The aims of the study were to attempt to answer the following questions; what proportion of women know how to and are able to exercise their pelvic floor and for those who cannot can they be trained and motivated to do so. This was a nested design comprising a prospective cohort study together with a controlled trial intervention after baseline assessment in the cohort study for a defined at-risk group.

ELIGIBILITY:
Inclusion Criteria:

Able to give consent Aged above 18 years modified Oxford score, MOS, ≤ 2

Exclusion Criteria:

Unable to give consent

-

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2002-04; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
maximal vaginal squeeze pressure (perineometry). | monthly for 3 months

SECONDARY OUTCOMES:
endurance of contraction (perineometry)and digital vaginal palpation (MOS). | monthly for 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Robert Freeman, MD, Principal Investigator — University Hospital Plymouth NHS Trust
Locations (1):
- Plymouth Hospitals NHS Trust, Plymouth, Devon, United Kingdom

REFERENCES:
- [Derived] Waterfield A, Waterfield M, Campbell J, Freeman R. Can effective supervised pelvic floor muscle training be provided by primary care nurses? A randomized controlled trial. Int Urogynecol J. 2021 Oct;32(10):2717-2725. doi: 10.1007/s00192-021-04692-3. Epub 2021 Feb 23. PMID 33624122